CLINICAL TRIAL: NCT05452733
Title: Toward a Real-time Access to Sleepers' Mental Content
Acronym: SleepDance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of personnel to perform the tests
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP220764
Record Dates: First submitted 2022-06-17; First posted 2022-07-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Memory Reactivation; Memory Consolidation; Sleepwalking
Keywords: sleepwalking; sleep; memory consolidation; reactivation; dream; targeted memory reactivation
MeSH Terms: conditions — Somnambulism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleepwalking patient (Experimental)
  Interventions: Behavioral: differences of behavior between sleepwalking and non sleepwalking patient
- Non sleepwalking patient (Active Comparator)
  Interventions: Behavioral: differences of behavior between sleepwalking and non sleepwalking patient

INTERVENTIONS:
Behavioral: differences of behavior between sleepwalking and non sleepwalking patient — movement registry done by camera when low intensity sound are send to patient during sleep.

SUMMARY:
Sleep is crucial for global cognitive functioning, but its exact functions and mechanisms are still poorly understood. Cognitive studies of sleep typically rely on linking electrophysiological changes measured during sleep with behavioral and neural changes collected in tasks performed during wakefulness. What concomitantly happens in the mind of sleeping subjects is often ignored, certainly because it is virtually inaccessible. Yet, major advances in the understanding of human behaviors have resulted from an integrated approach that combines both neural and cognitive measures of their ongoing mental processes. The goal of this study is to provide real-time measures of the cognitive processes occurring within sleep.

To prompt real-time access to the sleeping mind, investigators will use auditory stimulation in people with unique sleep peculiarities: sleepwalkers whose overt behaviours may enable to objectively visualize ongoing cognitive processes during non-REM (NREM) sleep.

DETAILED DESCRIPTION:
Investigators aim to offer a quantifiable, real-time measure of memory processing during NREM sleep by using memory-related cues to influence which behaviours sleepwalkers will exhibit. Because sleepwalking is characterized by complex behaviors emerging from NREM sleep, it could provide an observable window into mental activity in NREM sleep. While neuronal memory reactivations have largely been demonstrated in sleeping rodents, evidence for the existence of such reactivations in humans is at best indirect. Here, investigators will use targeted memory reactivation (TMR), a tool that allows to control which individual memories are reactivated on a trial by trial basis. TMR consists in associating sensory cues with a specific learning, then re-applying these cues during subsequent sleep to trigger the reactivation of the corresponding learning. Sleepwalkers will be trained on a modified version of the serial reaction time task: sleepwalkers will perform as fast and accurately as possible a sequence of gestures in response to auditory cues. Investigators goals are to: i) show that playing the auditory cues during NREM sleep triggers a behavioral replay of the learned 'choreography' in sleepwalkers, ii) quantify, with a gesture recognition algorithm, how the sleep gestures differ from the wake ones (speed, accuracy, sequence fidelity), and iii) test whether this evoked replay is accompanied by a congruent dream.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-35 y.o
* Written consent
* Affiliated to social security
* Sleepwalking (group patients only)

Exclusion Criteria:

* Psychiatric or neurologic disorder
* Sleep disorder except sleepwalking for the patient group
* Surdity
* Pain or physical disability affecting the upper limbs
* Consumption of drugs altering sleep structure
* Subjects under legal protection

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Behavioral reaction | 2 days
  number of behavioral reactivations of the motor sequence following the auditory cues during sleep

SECONDARY OUTCOMES:
Evaluation of targeted memory reactivation (TMR) success in sleepwalkers by movements test | 2 days
  test whether performance is better for movements that have been cued during sleep (vs. uncued ones) in sleepwalkers
Quantification of movements exhibited during sleep | 2 days
  The quantification of movement will be evaluated by combinaison of the reaction time, speed and precision of movements exhibited by sleepwalkers during sleep vs. wakefulness
Determination of the link between dream and sensory cues | 2 days
  Comparison between the number of dreams related to the motor sequence on the 2nd night (after TMR) vs. during the 1st one.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Arnulf, MD PhD, Principal Investigator — APHP; Delphine Oudiette, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Service des Pathologies du Sommeil, Hôpital Pitié-Salpétrière, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided